CLINICAL TRIAL: NCT04172428
Title: Comparison of Compact 3T, Conventional 3T, and 7T Scanners Using Task Based and Resting State fMRI
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, David F. Black, Principal Investigator, Mayo Clinic
Other Study IDs: 19-004228
Record Dates: First submitted 2019-09-05; First posted 2019-11-21 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy volunteers: Young healthy volunteers between the ages of 18-55.
  Interventions: Diagnostic Test: Functional MRI (fMRI)

INTERVENTIONS:
Diagnostic Test: Functional MRI (fMRI) — fMRI will be done on 3 separate MRI scanners to compare.

SUMMARY:
Comparison of 3 MRI scanners.

DETAILED DESCRIPTION:
Comparing the strengths and weaknesses of 3 different MRI scanners in their performance of a functional MRI (an MRI that shows which areas in the brain are active during some sort of task).

ELIGIBILITY:
Inclusion Criteria:

1) Men and Women aged 18-55

Exclusion Criteria:

1. Patients with safety contraindications to MRI scanning at 3T.
2. Patients unable to adequately perform the fMRI task due to physical, neurological, or cognitive disability.
3. Patients that demonstrate 3 mm or greater translational head motion during scanning of the fMRI rhyming task data sets.
4. Pregnant women.
5. Patients that have implanted medical devices or other safety contraindications for a 7T or 3T MRI exam.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young healthy volunteers ages 18-55, English must be primary language
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Statistical maxima of fMRI language and motor area activations. | Approximately 6 months after last subject is scanned
  For the task-based fMRI comparison, a region of interest will be drawn around activation maps overlying Broca's and Wernicke's language areas as well as the hand motor area. The data regarding each of the three regions will be treated separately. The statistical maxima for functional activation within these areas will be measured and compared using the same areas and technique on the three scanner platforms to determine which is the highest. This will be performed using the PRISM software we already use clinically to interpret fMRI.
Signal to noise ratio assessment of resting state. | Approximately 6 months after last subject is scanned
  For the resting state fMRI comparison, a standard measurement of signal to noise ratio will be employed specifically using the default mode network. This data will be reported separately from the task based outcome #1 as they are unrelated. Because this is a ratio is has no units of measurement.

SECONDARY OUTCOMES:
Neuroradiologist preference for scanner array. | Approximately 6 months after last subject is scanned
  Two board certified neuroradiologists will simply rank the 3 different scanner platforms (3T, Compact 3T, or the 7T) from most to least preferred for interpreting language and motor task-based fMRI's. This will be their overall qualitative gestalt based on years of daily experience reading these types of studies.

CONTACTS AND LOCATIONS:
Overall Officials: David F Black, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials